CLINICAL TRIAL: NCT05902169
Title: A Randomized, Open-label, Multicentric, Two-arm Pivotal Trial of SonoCloud-9 Combined With Carboplatin (CBDCA) vs Standard of Care Lomustine (CCNU) or Temozolomide (TMZ) in Patients Undergoing Planned Resection for First Recurrence Glioblastoma.
Brief Title: Sonocloud-9 in Association With Carboplatin Versus Standard-of-Care Chemotherapies (CCNU or TMZ) in Recurrent GBM
Acronym: SONOBIRD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CarThera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC9-GBM-03; 2023-505829-14-00 (Other: EU CT Number)
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; GBM
Keywords: carboplatin; SonoCloud; blood-brain barrier; Low Intensity Pulsed Ultrasound (LIPU)
MeSH Terms: conditions — Glioblastoma | interventions — Carboplatin; Lomustine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: SonoCloud-9 Ultrasound + Carboplatin (Experimental): The SonoCloud-9 (SC9) device will be implanted in the skull bone window upon completion of tumor resection and routine craniotomy. Carboplatin (CBDCA) will be administered intravenously prior to sonication. The CBDCA/SC9 treatment will be repeated every 3 weeks (depending on patient's tolerability) until disease progression or as clinically indicated. Administration of up to 7 cycles is planned.
  Interventions: Device: SonoCloud-9 (SC9); Drug: Carboplatin
- Control Arm: SoC single agent chemotherapy TMZ or CCNU (Active Comparator): Standard of Care (SoC) treatment with either temozolomide (TMZ) or lomustine (CCNU).
  Standard TMZ chemotherapy as a single oral dose every 4 weeks for up to 6 cycles.
  Standard CCNU chemotherapy as a single oral dose every 6 weeks for up to 4 cycles.
  Interventions: Drug: Lomustine; Drug: Temozolomide

INTERVENTIONS:
Device: SonoCloud-9 (SC9) — Implantation of SC9 device and repeat activation at constant acoustic pressure
  Arms: Experimental Arm: SonoCloud-9 Ultrasound + Carboplatin
Drug: Carboplatin — Dose of carboplatin AUC 5 mg/ml.min-1 calculated using Calvert's formula:
  Dose (mg) = target AUC (mg/mL x minute) x [glomerular filtration rate (GFR) mL/minute + 25].
  Other Names: CycloButane DiCarboxylic Acid (CBDCA)
  Arms: Experimental Arm: SonoCloud-9 Ultrasound + Carboplatin
Drug: Lomustine — Dosed and administered per labelling.
  Other Names: 1-(2-chloroethyl)-3-cyclohexyl-1-nitrosourea (CCNU)
  Arms: Control Arm: SoC single agent chemotherapy TMZ or CCNU
Drug: Temozolomide — Dosed and administered per labelling.
  Other Names: Temodal
  Arms: Control Arm: SoC single agent chemotherapy TMZ or CCNU

SUMMARY:
The brain is protected from any toxic or inflammatory molecule by the blood-brain barrier (BBB). This physical barrier is located at the level of the blood vessel walls. Because of these barrier properties, the blood vessels are also impermeable to the passage of therapeutic molecules from the blood to the brain. The development of effective treatments against glioblastoma is thus limited due to the BBB that prevents most drugs injected in the bloodstream from getting into brain tissue where the tumour is seated. The SonoCloud-9 (SC9) is an investigational device using ultrasound technology and specially developed to open the BBB in the area of and surrounding the tumour. The transient opening of the BBB allows more drugs to reach the brain tumour tissue. Carboplatin is a chemotherapy that is approved to treat different cancer types alone or in combination with other drugs, and has been used in the treatment of glioblastoma. Despite its proven efficacy in the laboratory on glioblastoma cells, carboplatin does not readily cross the BBB in humans. A clinical trial has shown that in combination with the SonoCloud-9, more carboplatin can reach the brain tumour tissue. The objective of the proposed trial is to show that the association - carboplatin with the SonoCloud-9 - will increase efficacy of the drug in patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven glioblastoma (WHO criteria 2021), absence of IDH mutation demonstrated by negative IDH1 R132H staining on Immunohistochemistry.
2. Patient must have received prior first line therapy that must have contained both:

   1. Prior surgery or biopsy and standard fractionated radiotherapy (1.8-2 Gy/fraction, >56 Gy<66 Gy) or hypofractionated radiotherapy (15 x 2.66 Gy or similar regimen)
   2. One line of maintenance chemotherapy and/or immune- or biological therapy, (with or without Tumor-Treating Fields)
3. First, unequivocal disease progression with

   1. measurable tumor (>100 mm2 or 1 cm3, based on RANO criteria) documented (e.g., increase of 25% in tumor diameter) on MRI performed within 14 days of inclusion and,
   2. interval of a minimum of 12 weeks since the completion of prior radiotherapy, unless there is a new lesion outside the radiation field or unequivocal evidence of viable tumor on histopathological sampling
4. Patient is candidate for craniotomy and at least 50% resection of enhancing region
5. Maximal enhancing tumor diameter prior to inclusion ≤ 5 cm on T1w. (In case of planned lobectomy, post operative peritumoral brain or residual size ≤5 cm)
6. WHO performance status ≤ 2 (equivalent to Karnofsky Performance Status (KPS) ≥ 70)
7. Age ≥ 18 years
8. Participant must be recovered from acute toxic effects (<grade 2) of all prior anticancer therapy. Interval since last therapy to presumed date of surgery of at least:

   1. ≥ 4 weeks or 5 half-lives (whichever is shorter) for

      * Cytotoxic
      * Other small chemical entity (e.g., targeted therapy)
      * For biologics (e.g., antibodies, except bevacizumab)
   2. ≥ 6 weeks of prior bevacizumab
9. Adequate hematologic, hepatic, and renal laboratory values within 14 days of inclusion i.e.:

   1. Hemoglobin ≥ 10 g/dL, platelets ≥ 100,000/mm3, neutrophils ≥ 1500/mm3.
   2. Liver function test with ≤ grade 1 alterations, except if due to antiepileptic drug therapy or isolated increased bilirubin due to Gilbert syndrome
   3. Estimated glomerular filtration rate (eGFR) of at least 60 mL/min/1.73 m2 using Cockcroft Gault formula
10. Patient able to understand clinical trial information and willing to provide signed and informed consent
11. Patient of childbearing potential must have a negative pregnancy test within 14 days of inclusion and must agree to use a medically-acceptable method of birth control during the treatment period and, if randomized in the experimental arm, for at least 1 month after the last cycle of carboplatin
12. A male patient must agree to use condoms during the treatment period and, if randomized in the experimental arm, for at least 3 months after the last cycle of carboplatin; the patient must also refrain from donating sperm during this period.
13. Patient must be a beneficiary of a health plan that covers routine patient care costs. Patient must be a beneficiary of or affiliated with a social security scheme (according to country-specific requirements)

Non-Inclusion Criteria:

1. Multifocal enhancing tumor on T1w (unless all localized in a 5 cm diameter area)
2. Posterior fossa tumor
3. Known BRAF/ NTKR mutated patients
4. Patient at risk of surgery site infection (e.g., 2 or more previous craniotomies/neurosurgery within the last 3 months, poor skin condition, and/or previously infected surgical field, or any other condition that is of increased infectious risk in the opinion of the neurosurgeon)
5. Patient treated at high, stable -or average- dose of corticosteroids (≥ 6 mg/day dexamethasone or equivalent) in the 7 days prior to inclusion. Patients on dexamethasone for reasons other than mass effect may still be enrolled.
6. Contra-indication to carboplatin, CCNU or TMZ
7. Known history of hypersensitivity reactions to perflutren lipid microsphere components or to any of the inactive ingredients in ultrasound resonator
8. Patient has received bevacizumab for other reasons (such as tumor progression) than treating edema
9. Peripheral neuropathy or neuropathy ≥ grade 2
10. Uncontrolled epilepsy or evidence of intracranial pressure
11. Patient with known intracranial aneurism or having presented intra-tumor significant spontaneous hemorrhage
12. Patient with unremovable coils, clips, shunts, intravascular stents, and/or wafer, or reservoirs
13. Patient with medical need to be on continued anti-platelet aggregation therapy and/or anticoagulation. Patients for whom anticoagulation/platelet aggregation can be temporarily interrupted may be eligible after discussion and prior authorization by the sponsor.
14. Patient receiving enzyme-inducing antiepileptic drugs (namely phenytoin, carbamazepine and derivatives, phenobarbital), unless switched on another antiepileptic regimen
15. History of other malignancy within 3 years prior to study start with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma, non-melanomatous skin cancer or carcinoma in situ of the uterine cervix
16. Patient with known or suspected active or chronic infections
17. Patient with known significant cardiac disease, known to have right-to-left shunts, severe pulmonary hypertension (pulmonary artery pressure > 90 mm Hg), uncontrolled systemic hypertension, or acute respiratory distress syndrome
18. Known sensitivity/allergy to gadolinium, or other intravascular contrast agents
19. Patient with impaired thermo-regulation or temperature sensation
20. Pregnant, or breastfeeding patient
21. Any other serious patient medical or psychological condition that may interfere with adequate and safe delivery of treatment and care (e.g., positive human immunodeficiency virus [HIV] status, potential blood-borne infections,…), circumstance (e.g., sinus opening during surgery), psychological, morphological characteristics (e.g., skin characteristics, bone thickness), or any pre-existing comorbidities that in the investigator's opinion may prevent the implantation of the device, may impair the ability of the patient to receive treatment with SonoCloud-9 or may be confounding for evaluation of the clinical trial endpoints
22. Patients under guardianship, curatorship, under legal protection or deprived of liberty by an administrative or judicial decision

Exclusion Criterion:

Occurrence of any major medical illnesses or impairments that in the Investigator's opinion may hampered the ability of the patient to receive treatment with SonoCloud-9 or may be confounding for evaluation of the clinical endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2028-01-28 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 24 months
  Survival status will be collected during the treatment period, for up to 7 months (short-term follow-up) and then every 3 months as standard of care follow-up (long-term follow-up) until participant's 'End of Study', defined as end of survival follow-up period, death, withdrawal of consent for the collection of data, or 'lost to follow-up' (whichever comes first).

SECONDARY OUTCOMES:
Tumor Growth Rate | Up to week 24
  Tumor Growth Rate will be determined by measuring hyperintense tumor volume using T1w contrast-enhancing tumor-related region from post-surgery MRI baseline to unequivocal progression MRI (i.e., suspected radiologic progression confirmed by repeat scan).
Progression Free Survival (PFS) | Up to 24 months
  Defined as the time from date of randomization to the earlier of the following events: unequivocal tumor progression as determined by IRC per RANO criteria or death due to any cause.
Overall survival at 12 months (OS12) | 12 months
  Defined as the proportion of participants alive at 12 months
Overall survival at 18 months (OS18) | 18 months
  Defined as the proportion of participants alive at 18 months
Progression-free survival at 6 months (PFS6) | 6 months
  Defined as the proportion of participants without disease progression or death due to any cause at 6 months.

OTHER OUTCOMES:
Safety and Tolerability | Up to week 24
  Frequency and severity of adverse events scored according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, from surgery to End-of-Trial Intervention visit

CONTACTS AND LOCATIONS:
Locations (48):
- United States (19):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - UCHealth, Aurora, Colorado
  - Mayo Clinic of Jacksonville Florida, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Weill Cornell Medicine, New York, New York
  - NewYork-Presbyterian / Columbia University Irving Medical Center, New York, New York
  - Lennox Hill Hospital, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Houston Health Science Center, Houston, Texas
  - University of Utah, Hunstman Cancer Institute, Salt Lake City, Utah
- Medizinische Universitaet Innsbruck, Innsbruck, Austria
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
  - CHU de Liège, Liège
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- France (4):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Hôpital de La Timone, Marseille
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Foch, Suresnes
- Germany (5):
  - Charité Universitätsmedizin Berlin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Neurochirurgie uniklinik Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Essen Klinik für Neurologie, Essen
- Italy (5):
  - Ospedale Bellaria, Bologna
  - Ospedale Civile di Livorno, Livorno
  - Istituto Oncologico Veneto, Padua
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliero Universitaria Città della Salute e della Scienza di Torino, Torino
- Netherlands (2):
  - Erasmus Medisch Centrum (Erasmus MC), Rotterdam
  - Haaglanden Medisch Centrum, The Hague
- Spain (5):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Switzerland (2):
  - Inselspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpentier A, Canney M, Vignot A, Reina V, Beccaria K, Horodyckid C, Karachi C, Leclercq D, Lafon C, Chapelon JY, Capelle L, Cornu P, Sanson M, Hoang-Xuan K, Delattre JY, Idbaih A. Clinical trial of blood-brain barrier disruption by pulsed ultrasound. Sci Transl Med. 2016 Jun 15;8(343):343re2. doi: 10.1126/scitranslmed.aaf6086. PMID 27306666
- [Background] Sonabend AM, Gould A, Amidei C, Ward R, Schmidt KA, Zhang DY, Gomez C, Bebawy JF, Liu BP, Bouchoux G, Desseaux C, Helenowski IB, Lukas RV, Dixit K, Kumthekar P, Arrieta VA, Lesniak MS, Carpentier A, Zhang H, Muzzio M, Canney M, Stupp R. Repeated blood-brain barrier opening with an implantable ultrasound device for delivery of albumin-bound paclitaxel in patients with recurrent glioblastoma: a phase 1 trial. Lancet Oncol. 2023 May;24(5):509-522. doi: 10.1016/S1470-2045(23)00112-2. PMID 37142373
- See also: CARTHERA — http://www.carthera.eu